CLINICAL TRIAL: NCT02690025
Title: A Phase 2 Trial Testing ZP1848 in Patients With SBS
Acronym: glepaglutide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Collaborators: Larix A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZP1848-15073
Record Dates: First submitted 2016-02-12; First posted 2016-02-24 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ZP1848 High dose (Experimental): s.c. administration of high dose
  Interventions: Drug: ZP1848
- ZP1848 Medium dose (Experimental): s.c. administration of medium dose
  Interventions: Drug: ZP1848
- ZP1848 Low dose (Experimental): s.c. administration of low dose
  Interventions: Drug: ZP1848

INTERVENTIONS:
Drug: ZP1848

SUMMARY:
A proof-of-concept, dose finding, controlled, single-center, randomized, double-blind, fixed dose phase 2 trial with ZP1848 in patients with Short Bowel Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Following receipt of verbal and written information about the trial, the patient must provide signed informed consent before any trial related activity is carried out.
* Age ≥ 18 years and ≤ 90 years
* Stable SBS patients with intestinal insufficiency or failure, where the last surgical resection of gut tissue was performed at least 1 year ago
* A stable PS volume ( < 25% change in volume or energy content) for four weeks prior to randomization for patients requiring PS
* Wet weight of fecal excretion ≥ 1500 g/day demonstrated during a hospital stay prior to screening or during at least one day of the first baseline balance study.
* Stable body weight (<5% weight deviance in the three months prior to screening)

Exclusion Criteria:

* Patients with known or suspected intestinal strictures of clinical relevance as judged by the Investigator
* Active inflammatory bowel disease (IBD) or fistula during the screening period as judged by conventional means of the Investigator.
* Crohn's disease patients not being in clinical remission for the last 12 weeks prior to randomization
* Cardiac disease defined as: Decompensated heart failure (NYHA class III-IV) and/or diagnosis of unstable angina pectoris and/or myocardial infarction within the last 6 months prior to screening
* History of cancer (except resected cutaneous basal or squamous cell carcinoma and except in situ cervical cancer) unless it can be documented that the patient has been in a disease-free state for at least 5 years (except colon cancer: patients with a history of colon cancer generally have to be excluded)
* eGFR (by the MDRD formula) <30 mL/min/1.73 m2
* Clinically meaningful renal disease as judged by the Investigator

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-02; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
The Primary endpoint is the absolute change from baseline to the end of three week treatment periods of wet weight of ostomy output or diarrhea measured separately over each of the two treatment periods. | 3 weeks

SECONDARY OUTCOMES:
Relative change from baseline to the end of treatment of wet weight of ostomy output or diarrhea measured separately over each of the two treatment periods | 3 weeks
Absolute change from baseline to the end of treatment of urine weight measured separately over each of the two treatment periods | 3 weeks
Relative change from baseline to the end of treatment of urine weight measured separately over each of the two treatment periods | 3 weeks
Absolute change from baseline to the end of treatment of wet weight absorption measured separately over each of the two treatment periods | 3 weeks
Relative change from baseline to the end of treatment of wet weight absorption measured separately over each of the two treatment periods | 3 weeks
Absolute change from baseline to the end of treatment of the intestinal absorption of electrolytes measured separately over each of the two treatment periods | 3 weeks
Relative change from baseline to the end of treatment of the intestinal absorption of electrolytes measured separately over each of the two treatment periods | 3 weeks
Absolute change from baseline to the end of treatment of the intestinal absorption of macronutrients measured separately over each of the two treatment periods | 3 weeks
Relative change from baseline to the end of treatment of the intestinal absorption of macronutrients measured separately over each of the two treatment periods | 3 weeks
Change in SF-36 score | 3 weeks
Incidence of Adverse Events | 15 weeks
Incidence of Anti Drug Antibodies | 15 weeks
Absolute change from baseline to the end of treatment of urine weight minus oral intake measured separately over each of the two treatment periods | 3 weeks
Relative change from baseline to the end of treatment of urine weight minus oral intake measured separately over each of the two treatment periods | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gertrud Koefoed Rasmussen, MSc, Study Director — Zealand Pharma A/S
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hvistendahl MK, Naimi RM, Hansen SH, Rehfeld JF, Kissow H, Pedersen J, Dragsted LO, Sonne DP, Knop FK, Jeppesen PB. Bile acid-farnesoid X receptor-fibroblast growth factor 19 axis in patients with short bowel syndrome: The randomized, glepaglutide phase 2 trial. JPEN J Parenter Enteral Nutr. 2022 May;46(4):923-935. doi: 10.1002/jpen.2224. Epub 2021 Sep 1. PMID 34287979
- [Derived] Naimi RM, Hvistendahl M, Nerup N, Ambrus R, Achiam MP, Svendsen LB, Gronbaek H, Moller HJ, Vilstrup H, Steensberg A, Jeppesen PB. Effects of glepaglutide, a novel long-acting glucagon-like peptide-2 analogue, on markers of liver status in patients with short bowel syndrome: findings from a randomised phase 2 trial. EBioMedicine. 2019 Aug;46:444-451. doi: 10.1016/j.ebiom.2019.07.016. Epub 2019 Jul 17. PMID 31326433
- [Derived] Naimi RM, Hvistendahl M, Enevoldsen LH, Madsen JL, Fuglsang S, Poulsen SS, Kissow H, Pedersen J, Nerup N, Ambrus R, Achiam MP, Svendsen LB, Holst JJ, Hartmann B, Hansen SH, Dragsted LO, Steensberg A, Mouritzen U, Hansen MB, Jeppesen PB. Glepaglutide, a novel long-acting glucagon-like peptide-2 analogue, for patients with short bowel syndrome: a randomised phase 2 trial. Lancet Gastroenterol Hepatol. 2019 May;4(5):354-363. doi: 10.1016/S2468-1253(19)30077-9. Epub 2019 Mar 15. PMID 30880176